CLINICAL TRIAL: NCT04620213
Title: Randomized, Parallel Arm, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically-Induced Mydriasis in Healthy Subjects
Brief Title: Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically-Induced Mydriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXRM-301 (MIRA-2)
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Mydriasis; Dilation
Keywords: Nyxol; Pharmacologically Induced Mydriasis; Dilation
MeSH Terms: conditions — Mydriasis; Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Ophthalmic Solution 0.75% (Experimental): 2 drops in study eye and 1 drop in non-study eye, 1 hour post pharmacologically-induced mydriasis
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%
- Phentolamine Ophthalmic Solution Vehicle (Placebo Comparator): 2 drops in study eye and 1 drop in non-study eye, 1 hour post pharmacologically-induced mydriasis
  Interventions: Other: Phentolamine Ophthalmic Solution Vehicle (Placebo)

INTERVENTIONS:
Drug: Phentolamine Ophthalmic Solution 0.75% — 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol; Nyxol®
  Arms: Phentolamine Ophthalmic Solution 0.75%
Other: Phentolamine Ophthalmic Solution Vehicle (Placebo) — Topical sterile ophthalmic solution
  Arms: Phentolamine Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of Nyxol to expedite the reversal of pharmacologically-induced mydriasis across multiple mydriatic agents with an emphasis on phenylephrine
* To evaluate the efficacy of Nyxol to return subjects to baseline accommodation after worsening (with cycloplegic agents tropicamide and Paremyd)
* To evaluate the safety of Nyxol
* To evaluate any additional benefits of the reversal of pharmacologically-induced mydriasis

DETAILED DESCRIPTION:
A randomized, parallel arm, double-masked, placebo-controlled Phase 3 study in at least 168 randomized subjects (160 completed), evaluating the safety and efficacy of Nyxol in subjects with pharmacologically-induced mydriasis.

Following the successful completion of screening, each subject will be stratified by eye color and then simultaneously be randomized to mydriatic agent (unmasked) and treatment (masked).

Treatment randomization will be 1:1, Nyxol or placebo (vehicle).

Stratification by iris color will be 1:1, light or dark irides.

The mydriatic agent randomization will be 3:1:1 (2.5% phenylephrine, 1% tropicamide, and Paremyd). That is, approximately 60% of the randomized subjects will receive one drop of 2.5% phenylephrine 1 hour before treatment (96 completed subjects), approximately 20% will receive one drop of 1% tropicamide 1 hour before treatment (32 completed subjects), and approximately 20% will receive Paremyd 1 hour before treatment (32 completed subjects).

At the treatment visit, subjects who have been randomized and stratified by iris color (1:1 [light/dark]) will receive one of three approved mydriatic agents approximately 1 hour prior to receiving study treatment. Measurements will be measured before (-1 hour /baseline) and 60 minutes after (maximum/0 minutes) the mydriatic agent instillation in each eye (i.e. right before the study treatment is administered), and at 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, and 6 hours after treatment dosing. Measurements will include pupil diameter (PD), distance and near visual acuity (VA), accommodation, and redness in each eye.

At the Follow-Up Visit, which is 1 day after Visit 1, measurements will again be recorded 24 hours after treatment dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 12 years of age
2. Otherwise healthy and well controlled subjects

Exclusion Criteria:

Ophthalmic (in either eye):

1. Clinically significant ocular disease as deemed by the Investigator that might interfere with the study
2. Unwilling or unable to discontinue use of contact lenses at screening until study completion
3. Unwilling or unable to suspend use of topical medication at screening until study completion
4. Ocular trauma, ocular surgery or non-refractive laser treatment within the 6 months prior to screening
5. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind within 7 days of screening
6. Recent or current evidence of ocular infection or inflammation in either eye
7. History of diabetic retinopathy or diabetic macular edema
8. Closed or very narrow angles that in the Investigator's opinion are potentially occludable if the subject's pupil is dilated
9. History of any traumatic (surgical or nonsurgical) or non-traumatic condition affecting the pupil or iris
10. Known allergy or contraindication to any component of the mydriatic agents or the vehicle formulation
11. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal

Systemic:

1. Known hypersensitivity or contraindication to α- and/or β adrenoceptor antagonists.
2. Clinically significant systemic disease that might interfere with the study
3. Initiation of treatment with or any changes to the current dosage, drug or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to screening, or during the study
4. Participation in any investigational study within 30 days prior to screening
5. Females of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control
6. Resting HR outside the normal range (50-110 beats per minute)
7. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Clinical Site 11, Newport Beach, California
  - Clinical Site 10, San Diego, California
  - Clinical Site 9, Longwood, Florida
  - Clinical Site 6, Orlando, Florida
  - Clinical Site 2, Roswell, Georgia
  - Clinical Site 7, Pittsburg, Kansas
  - Clinical Site 3, Shawnee Mission, Kansas
  - Clinical Site 5, Athens, Ohio
  - Clinical Site 12, Cincinnati, Ohio
  - Clinical Site 1, Cleveland, Ohio
  - Clinical Site 8, Warwick, Rhode Island
  - Clinical Site 4, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Started | 94 | 91
Completed | 94 | 91
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (14.04) | 32.8 (13.55) | 33.4 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 113
  Male | 36 | 36 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 74 | 144
  American Indian or Alaska Native | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 16 | 33
  Asian | 6 | 3 | 9
Irides Type: Light, Dark [Count of Participants; unit: Participants]
  Light | 45 | 45 | 90
  Dark | 49 | 46 | 95
Mydriatic Agent [Count of Participants; unit: Participants]
  Phenylephrine | 56 | 55 | 111
  Tropicamide | 19 | 18 | 37
  Paremyd | 19 | 18 | 37
Baseline Pupil Diameter (Study Eye) [Mean (Standard Deviation); unit: mm] | 5.085 (0.9295) | 5.177 (0.9678) | 5.130 (0.9471)
Baseline Accomodation (Study Eye) [Mean (Standard Deviation); unit: D] | 10.47 (20.373) | 8.25 (5.230) | 9.38 (14.980)
Baseline BCDVA (Study Eye) [Mean (Standard Deviation); unit: Letters] | 57.0 (4.10) | 58.6 (4.49) | 57.8 (4.36)
Baseline DCNVA [Mean (Standard Deviation); unit: Letters] | 65.6 (10.63) | 67.0 (9.74) | 66.3 (10.20)
Baseline IOP (Study Eye) [Mean (Standard Deviation); unit: mmHg] | 15.3 (2.78) | 15.1 (2.95) | 15.2 (2.85)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects' Study Eyes With Pupil Diameter Returning to Baseline
Description: Percentage of subjects' study eyes returning to less than or equal to 0.2 mm from baseline pupil diameter
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 94 | 91
Participants | 46 | 6

2. Secondary Outcome: Percent of Subjects' Study Eyes Pupil Diameter Returning to Baseline
Description: Percentage of subjects' study eyesreturning to less than or equal to 0.2 mm from baseline pupil diameter
Time Frame: up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 94 | 91
Participants
  30 minutes | 1 | 3
  60 minutes | 26 | 2
  90 minutes | 46 | 6
  2 hours | 55 | 10
  3 hours | 75 | 16
  4 hours | 77 | 27
  6 Hours | 85 | 41
  24 Hours | 86 | 60

3. Secondary Outcome: Pupil Diameter (Change From Max)
Description: Change (mm) from maximum pharmacologically-induced mydriatic pupil diameter (0 minutes)
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 94 | 91
millimeters
  Baseline (-1 Hour) | 5.085 (0.9295) | 5.177 (0.9678)
  0 minutes | 7.207 (1.024) | 7.197 (1.1717)
  30 minutes | 0.025 (0.4780) | 0.075 (0.4266)
  60 minutes | -1.308 (0.8705) | -0.122 (0.4055)
  90 minutes | -2.192 (1.0117) | -0.329 (0.4653)
  2 hours | -2.429 (0.9837) | -0.518 (0.5930)
  3 hours | -2.828 (0.9817) | -0.806 (0.6253)
  4 hours | -2.991 (1.0793) | -1.159 (0.8223)
  6 hours | -3.338 (1.0797) | -1.634 (1.0595)
  24 Hours | -3.375 (1.2302) | -2.173 (1.3868)

4. Secondary Outcome: Percent of Subjects With Unchanged Accommodation From Baseline
Description: Percentage of subjects with unchanged accommodation from baseline (-1 hour)
Time Frame: up to 6 hours
Population: Subjects within each overall treatment group were randomized to receive one of 3 mydriatic agents (3;1;1); therefore the number of subjects in the the subgroups do not match the overall number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 94 | 91
Participants
  Phenylephrine, 0 minutes: number analyzed (Participants) | 56 | 55
  Phenylephrine, 0 minutes: Unchanged from Baseline | 30 | 37
  Phenylephrine, 0 minutes: Changed from Baseline | 26 | 18
  Phenylephrine, 60 minutes: number analyzed (Participants) | 56 | 55
  Phenylephrine, 60 minutes: Unchanged from Baseline | 29 | 39
  Phenylephrine, 60 minutes: Changed from Baseline | 27 | 16
  Phenylephrine, 90 minutes: number analyzed (Participants) | 56 | 55
  Phenylephrine, 90 minutes: Unchanged from Baseline | 38 | 40
  Phenylephrine, 90 minutes: Changed from Baseline | 18 | 15
  Phenylephrine, 2 hours: number analyzed (Participants) | 56 | 55
  Phenylephrine, 2 hours: Unchanged from Baseline | 40 | 42
  Phenylephrine, 2 hours: Changed from Baseline | 16 | 13
  Phenylephrine, 3 hours: number analyzed (Participants) | 56 | 55
  Phenylephrine, 3 hours: Unchanged from Baseline | 38 | 45
  Phenylephrine, 3 hours: Changed from Baseline | 18 | 10
  Phenylephrine, 4 hours: number analyzed (Participants) | 56 | 55
  Phenylephrine, 4 hours: Unchanged from Baseline | 39 | 42
  Phenylephrine, 4 hours: Changed from Baseline | 17 | 13
  Phenylephrine, 6 hours: number analyzed (Participants) | 56 | 55
  Phenylephrine, 6 hours: Unchanged from Baseline | 43 | 48
  Phenylephrine, 6 hours: Changed from Baseline | 13 | 7
  Tropicamide, 0 Minutes: number analyzed (Participants) | 19 | 18
  Tropicamide, 0 Minutes: Unchanged from Baseline | 2 | 2
  Tropicamide, 0 Minutes: Changed from Baseline | 17 | 16
  Tropicamide, 60 Minutes: number analyzed (Participants) | 19 | 18
  Tropicamide, 60 Minutes: Unchanged from Baseline | 6 | 5
  Tropicamide, 60 Minutes: Changed from Baseline | 13 | 13
  Tropicamide, 90 Minutes: number analyzed (Participants) | 19 | 18
  Tropicamide, 90 Minutes: Unchanged from Baseline | 10 | 5
  Tropicamide, 90 Minutes: Changed from Baseline | 9 | 13
  Tropicamide, 2 Hours: number analyzed (Participants) | 19 | 18
  Tropicamide, 2 Hours: Unchanged from Baseline | 12 | 6
  Tropicamide, 2 Hours: Changed from Baseline | 7 | 12
  Tropicamide, 3 Hours: number analyzed (Participants) | 19 | 18
  Tropicamide, 3 Hours: Unchanged from Baseline | 13 | 8
  Tropicamide, 3 Hours: Changed from Baseline | 6 | 10
  Tropicamide, 4 Hours: number analyzed (Participants) | 19 | 18
  Tropicamide, 4 Hours: Unchanged from Baseline | 14 | 10
  Tropicamide, 4 Hours: Changed from Baseline | 5 | 8
  Tropicamide, 6 Hours: number analyzed (Participants) | 19 | 18
  Tropicamide, 6 Hours: Unchanged from Baseline | 14 | 12
  Tropicamide, 6 Hours: Changed from Baseline | 5 | 6
  Paremyd, 0 Minutes: number analyzed (Participants) | 19 | 18
  Paremyd, 0 Minutes: Unchanged from Baseline | 2 | 3
  Paremyd, 0 Minutes: Changed from Baseline | 17 | 15
  Paremyd, 60 Minutes: number analyzed (Participants) | 19 | 18
  Paremyd, 60 Minutes: Unchanged from Baseline | 6 | 6
  Paremyd, 60 Minutes: Changed from Baseline | 13 | 12
  Paremyd, 90 Minutes: number analyzed (Participants) | 19 | 18
  Paremyd, 90 Minutes: Unchanged from Baseline | 7 | 7
  Paremyd, 90 Minutes: Changed from Baseline | 12 | 11
  Paremyd, 2 Hours: number analyzed (Participants) | 19 | 18
  Paremyd, 2 Hours: Unchanged from Baseline | 9 | 7
  Paremyd, 2 Hours: Changed from Baseline | 10 | 11
  Paremyd, 3 Hours: number analyzed (Participants) | 19 | 18
  Paremyd, 3 Hours: Unchanged from Baseline | 11 | 10
  Paremyd, 3 Hours: Changed from Baseline | 8 | 8
  Paremyd, 4 Hours: number analyzed (Participants) | 19 | 18
  Paremyd, 4 Hours: Unchanged from Baseline | 14 | 11
  Paremyd, 4 Hours: Changed from Baseline | 5 | 7
  Paremyd, 6 Hours: number analyzed (Participants) | 19 | 18
  Paremyd, 6 Hours: Unchanged from Baseline | 14 | 11
  Paremyd, 6 Hours: Changed from Baseline | 5 | 7
  Tropicamide or Paremyd, 0 Minutes: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 0 Minutes: Unchanged from Baseline | 4 | 5
  Tropicamide or Paremyd, 0 Minutes: Changed from Baseline | 34 | 31
  Tropicamide or Paremyd, 60 Minutes: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 60 Minutes: Unchanged from Baseline | 12 | 11
  Tropicamide or Paremyd, 60 Minutes: Changed from Baseline | 26 | 25
  Tropicamide or Paremyd, 90 Minutes: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 90 Minutes: Unchanged from Baseline | 17 | 12
  Tropicamide or Paremyd, 90 Minutes: Changed from Baseline | 21 | 24
  Tropicamide or Paremyd, 2 Hours: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 2 Hours: Unchanged from Baseline | 21 | 13
  Tropicamide or Paremyd, 2 Hours: Changed from Baseline | 17 | 23
  Tropicamide or Paremyd, 3 Hours: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 3 Hours: Unchanged from Baseline | 24 | 18
  Tropicamide or Paremyd, 3 Hours: Changed from Baseline | 14 | 18
  Tropicamide or Paremyd, 4 Hours: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 4 Hours: Unchanged from Baseline | 28 | 21
  Tropicamide or Paremyd, 4 Hours: Changed from Baseline | 10 | 15
  Tropicamide or Paremyd, 6 Hours: number analyzed (Participants) | 38 | 36
  Tropicamide or Paremyd, 6 Hours: Unchanged from Baseline | 28 | 23
  Tropicamide or Paremyd, 6 Hours: Changed from Baseline | 10 | 13

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/91
Other Adverse Events (participants affected / at risk) | 48/94 | 8/91
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phentolamine Ophthalmic Solution 0.75% (N=94) | Phentolamine Ophthalmic Solution Vehicle (N=91)
Instillation site discomfort (General disorders) | 36 | 8
Conjunctival Hyperaemia (Eye disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT04620213/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT04620213/SAP_001.pdf